CLINICAL TRIAL: NCT02047435
Title: Integrating Lonely Elderly Patients in Workshops in a Cartoon Museum: An Efficacy Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Research Unit Of General Practice, Copenhagen (Other)
Collaborators: The Storm P. Museum (Unknown); University College Absalon (Other); EGV Foundation (Other); Danish Agency for Culture (Unknown)
Responsible Party: Principal Investigator, Frans Boch Waldorff, PhD, Research Unit Of General Practice, Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Storm-P-2014
Record Dates: First submitted 2014-01-24; First posted 2014-01-28 (Estimated); Last update posted 2014-05-23 (Estimated); Status verified 2014-01

CONDITIONS: Quality of Life; Social Isolation; Loneliness
Keywords: Social participation; Loneliness; General practice; Cultural institutions
MeSH Terms: conditions — Social Isolation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Information, event and workshops at a cartoon museum (Experimental)
  Interventions: Behavioral: Information, event and workshops at a cartoon museum
- Information and event at a cartoon museum (Active Comparator)
  Interventions: Behavioral: Information and event at a cartoon museum

INTERVENTIONS:
Behavioral: Information, event and workshops at a cartoon museum — 1. An event at the Storm P. Museum consisting of:
     * A guided tour at the museum
     * A representative from the municipal DaneAge Association will tell about the municipality's activities for the elderly.
     * The museum serves a refreshment and offer participants a season pass to the museum.
     And
  2. Workshops at The Storm P. museum, for up to 12 months with approximately two workshops a months. In collaboration with the museum the participants create memory material for nursing home resident with dementia. The workshop will use narrative as a method to give participants a mutual relationship that is perceived as meaningful and rewarding for each participant and in the dialogues a mutual understanding is created. The museum staff facilitates the process of storytelling using events, significant stories and artistic works by Storm P., to encourage the participants, via the method known as "narrative interview", to share similar stories from their life.
  Arms: Information, event and workshops at a cartoon museum
Behavioral: Information and event at a cartoon museum — 1. An event at the Storm P. Museum consisting of:
  * A guided tour at the museum
  * A representative from the municipal DaneAge Association will tell about the municipality's activities for the elderly.
  * The museum serves a refreshment and offer participants a season pass to the museum.
  Arms: Information and event at a cartoon museum

SUMMARY:
Social relationships are important to people and it affects their quality of life, morbidity and mortality.

This is a randomised controlled trial studying the effect of including older people with impaired social relationships and a perception of loneliness at workshops, at The Storm P. Museum - a museum about the well known Danish cartoonist Robert Storm Petersen.

The hypothesis is, that by including older lonely people with a impaired social participation in these workshops, they will increase the participants health related quality of life. The investigators also hypothesis, that the intervention will improve the participants perception of loneliness, social participation and physical function.

The intervention consist of a series of workshops at the Storm P. Museum. At these workshops the participants will create memory material for nursing home residents with dementia. The museum staff will facilitate a process of storytelling, using events, significant stories and artistic works by Storm P. and encourage the participants, by means of the "narrative interview" method to share similar stories from their life.

DETAILED DESCRIPTION:
Background:

Social relations are important to people and it affects their quality of life, morbidity and mortality. This is especially true among older people and social relations are also important for the management of chronic diseases. Those with strong social relations are less sick, and recover faster if they become sick. There is also a connection between social relations and death, as people with many social relations are more likely to live longer than people with few social relations. In Denmark it is assumed that poor social relationships causes between 1000-1500 deaths per year, equivalent to about 2% of all deaths.

This is a randomised controlled trial studying the effect of including older people with poor social relationships and a perception of loneliness at workshops, at The Storm P. Museum - a museum about the well known Danish cartoonist Robert Storm Petersen.

Hypothesis:

The hypothesis is, that by including older lonely people with a poor social participation in these workshops, they will increase the participants health related quality of life. The investigators also hypothesis, that the intervention will improve the participants perception of loneliness, social participation and physical function as well as mortality and nursing home placement at long term.

The intervention:

Both the intervention and the comparison group will be invited to an event at the Storm P. Museum.

This event consist of

* A guided tour of the collection with a presentation on Storm P. 's life and artistic work.
* A representative from the municipal DaneAge Association will subsequently tell about the municipality's activities for the elderly.
* The museum will serve a refreshment and offer participants a season pass to the museum.

In addition the intervention group will be invited to participate in a series of workshops at the Storm P. Museum with scheduled meetings twice a month. In collaboration with the museum, participants at these workshops will create memory material for nursing home residents with dementia.

The workshop will use narrative as a method to give participants a mutual relationship that is perceived as meaningful and rewarding for each participant. Storytelling is central in creating a cognitive, meaningful and holistic life. In our dialogues we create a mutual understanding. Stories are central to people and is used in making sense in transitions and essential decisions in your life.

The museum facilitates the process of storytelling using events, significant stories and artistic works by Storm P., and encourage the participants, via the method known as "narrative interview", to share similar stories from their life. This will not only benefit the participants, but also act as crucial empirical data collected via journal keeping for this project.

The intervention is planned to last for up to 12 months and outcome measures are collected at baseline, 9 months and at 18 months.

ELIGIBILITY:
Patients consulting their general practitioner in the municipality of Frederiksberg during february/Marts 2014. Who in a questionnaire have a low score of social participation and answers they often feel lonely.

The participants are allocated to the study consecutively.

Inclusion Criteria:

Age: 65 years or older, Consultation at the general practice during the project period, Impaired social participation and often/occasionally perceive loneliness, Provided written informed consent

Exclusion Criteria:

Do not talk or understand Danish, Terminal ill, Physically not able to participate, Low score on cognitive test (OMC test)

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-02; Primary Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Difference from baseline in summary Index of EuroQol -5D | Baseline, 9 months and 18 months
  Health related quality of life measured by EuroQol -5D

SECONDARY OUTCOMES:
Score of MMSE test | Baseline, 9 months, 18 months
  Score of Mini Mental State Examination (MMSE).
Score of GDS-15 items | baseline, 9 months and 18 months
  Score of the Geriatric Depression Scale (GDS)
"Timed up and go" test | Baseline, 9 months and 18 months
Consultation at general practice and hospital admission | Baseline, 9 months and 18 months
Score on Mobility-Tiredness scale | Baseline, 9 months and 18 months
Score on social participation scale | Baseline, 9 months and 18 months
  Based on three items. The analysis is made on the individual items as well as the total score
Loneliness | Baseline, 9 months and 18 months
  Based on an item with four categories.

OTHER OUTCOMES:
All cause mortality | 36 month
  A long term follow up analysis.
Permanent nursing home placement | 36 month
  Long term follow up analysis
Health economic analysis | 36 month

CONTACTS AND LOCATIONS:
Overall Officials: Frans B Waldorff, PhD, Principal Investigator — Research Unit Of General Practice, Copenhagen; Tina D Due, PhD student, Principal Investigator — Research Unit Of General Practice, Copenhagen
Locations (1):
- Research Unit of General Practice Copenhagen, Copenhagen, Denmark